CLINICAL TRIAL: NCT03974412
Title: Syncope Trial to Understand Tilt Testing Early or Recorders Study
Acronym: STUTTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00087832
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Syncope
Keywords: syncope; head-up tilt table; implantable loop recorder; pragmatic
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All eligible participants (Experimental): All eligible participants are randomly assigned to one of two interventions- early Head-Up Tilt Table procedure or early Implantable Loop Recorder. The assignment is random and at a 1:1 ratio between the two strategies.
  Interventions: Diagnostic Test: Head Up Tilt Table (HUT); Device: Implantable Loop Recorder

INTERVENTIONS:
Diagnostic Test: Head Up Tilt Table (HUT) — Participant randomized to open-label diagnostic strategy. Results and all follow-up care to be in the hands of treating cardiologist as this is a pragmatic study.
  the early HUT [protocol: supine pre-tilt phase 5 min, un-medicated HUT to 70 degrees for 20 minutes; if response negative then 400 μg of sublingual nitroglycerin and continued 70 degree tilt for 20 minutes]
Device: Implantable Loop Recorder — ILR is a small subcutaneously implanted device, lasting up to 3 years, that records heart rhythms, and which may be either auto-triggered or patientactivated.

SUMMARY:
Pragmatic research study to determine which of the two standard syncope therapies yields a faster path to diagnosis- head up tilt (HUT) table or implantable loop recorder (ILR).

DETAILED DESCRIPTION:
RESEARCH QUESTION: In syncope patients at least 50 years of age, a strategy of first conducting a tilt table (HUT) will provide an earlier diagnosis at less cost than a strategy of first implanting an implantable loop recorder (ILR).

BACKGROUND: Syncope is a common condition. Approximately 0.6%- 1.5% of all Emergency Department (ED) visits occurs for syncope and of these, anywhere from 12%-83% are admitted, depending on the country. The incidence rates for acute care visits increases with age and rises steeply after the age of 50 years. Approximately one third of patients have at least one recurrence of syncope in 3 years of follow-up. A recent analysis from Alberta found the total cost of syncope presentations to the ED was $530 million dollars over a 6-year period. Syncope has numerous causes, ranging from benign to life threatening, and determining the underlying etiology is often challenging. Reflex syncope (vasovagal) is the most frequent cause of syncope in all age groups and clinical settings. However, arrhythmic causes, with higher clinical risk, become more common in older patients, and are responsible for about 10% of syncope visits to the ED. The current approach for investigation of patients with unexplained syncope is usually unstructured, with multiple specialist evaluations, numerous and expensive tests, and recurring acute care visits. This results in high and unnecessary costs. There are three competing approaches to diagnosis: a structured history, head-up tilt (HUT) test, and implantable loop recorders (ILR).

Often syncope can be diagnosed on the basis of history, physical examination, and electrocardiogram (ECG). However, even after this initial evaluation, syncope may remain unexplained, accounting for as many as 41% of cases in older patients. In older patients, history is often less reliable, due to a lack of autonomic symptoms associated with vasovagal syncope, amnesia for pre-syncopal symptoms, and lack of witnesses. Further, co-morbidities and polypharmacy add complexity to the diagnostic process. HUT: The HUT test has been used to evaluate patients with syncope for nearly 3 decades. It is an orthostatic stress test to assess the susceptibility of a vasovagal response to a postural change from a supine to an upright position. A positive response is defined as inducible presyncope or syncope associated with hypotension, with or without bradycardia (including asystole) that reproduces clinical symptoms. HUT has been used in patients with suspected vasovagal syncope, when the history is unhelpful. Although enthusiasm has waned for the role of HUT in the evaluation of syncope due to variable protocols leading to high heterogeneity of test outcomes, false-positives in controls, and availability of long-term cardiac monitoring; there is good evidence for its usefulness.

ILR is a small subcutaneously implanted device, lasting up to 3 years, that records heart rhythms, and which may be either auto-triggered or patientactivated.

Early observational and case-control studies found that the ILR leads to earlier diagnosis and reduced the rate of unexplained syncope compared to HUT. Despite ILR entering routine clinic practice over the last 25 years, there are surprisingly few rigorous data of its use in the management of unexplained syncope. Comparisons of strategies of HUT and ILR: Two randomized controlled studies have reported on the diagnostic yield of an early ILR strategy compared to conventional testing including HUT in older patients with unexplained syncope. All reported an increased diagnostic accuracy with ILR and a lower cost per diagnosis, but each has substantial limitations. Study Structure: This will be a formal pragmatic study of 2 diagnostic strategies, designed around the PRECIS2 criteria addressing which test should be done first, and subsequent care will be left in the hands of the physician responsible for assessing syncope. Settings: Patients will be recruited from the ED, general cardiology, arrhythmia, and syncope clinics, and medical and cardiology wards.

Randomization: Patients will be randomized to either i) the early HUT [protocol:

supine pre-tilt phase 5 min, un-medicated HUT to 70 degrees for 20 minutes; if response negative then 400 μg of sublingual nitroglycerin and continued 70 degree tilt for 20 minutes] OR ii) early implant of ILR without hospital admission.

Regardless of the outcome, subsequent testing and care will be in the hands of the responsible physician. Patients will be seen 1 week after ILR implantation for wound assessment and to reinforce patient understanding of the activation process. Subsequent 3-year follow-up will occur according to the policies of the device clinic (usually every 6 months). Patients will be seen quickly after a symptomatic event.

ELIGIBILITY:
Inclusion Criteria:

* 50 years old
* syncope (defined in 2017 ACC/AHA/HRS guidelines[16]) in the prior 12 months
* diagnosis unclear after history, physical exam andelectrocardiogram
* no apparent risk of death due to the cause of syncope.

Exclusion Criteria:

* inability to give informed consent
* unable to attend routine follow up in device clinic
* positive carotid sinus massage.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis | 1 year
  the proportion of patients with a definite diagnosis by 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No